CLINICAL TRIAL: NCT07136519
Title: Toripalimab Plus Induction Chemotherapy Followed by Radiation Therapy Combined With Omega-3 for Locally Advanced Nasopharyngeal Carcinoma: A Phase II, Single Arm Clinical Trial
Brief Title: Toripalimab, Induction Chemotherapy, Radiation Therapy With Omega-3 for Locally Advanced Nasopharyngeal Carcinoma
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Affiliated Hospital of Guangdong Medical University (Other)
Responsible Party: Principal Investigator, Haiqing Luo, Director of Head and Neck Oncology Department, Affiliated Hospital of Guangdong Medical University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PJ2025-005
Record Dates: First submitted 2025-08-01; First posted 2025-08-22 (Actual); Last update posted 2025-08-22 (Actual); Status verified 2025-08

CONDITIONS: Nasopharyngeal Carcinoma (NPC)
Keywords: Toripalimab; Omega-3
MeSH Terms: conditions — Nasopharyngeal Carcinoma | interventions — toripalimab; Docosahexaenoic Acids; Radiotherapy; Taxes; Cisplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Toripalimab Plus Omega-3 (Experimental): Toripalimab Plus Induction Chemotherapy Followed by Radiation Therapy Combined with Omega-3
  Interventions: Drug: Toripalimab; Dietary Supplement: Omega-3; Radiation: radiotherapy; Drug: Paclitaxel (albumin bound); Drug: Cisplatin

INTERVENTIONS:
Drug: Toripalimab — 240mg Q3W
  Other Names: not have
Dietary Supplement: Omega-3 — During radiotherapy, take 6 capsules once a day
  Other Names: not have
Radiation: radiotherapy — radiotherapy
  Other Names: not have
Drug: Paclitaxel (albumin bound) — 260mg/m2 d1,Q3W
  Other Names: not have
Drug: Cisplatin — 80mg/m2 d2, Q3W
  Other Names: not have

SUMMARY:
The aim of this study is to evaluate the efficacy, adverse reactions, nutritional status analysis, and quality of life analysis of Toripalimab Plus Induction Chemotherapy Followed by Radiation Therapy Combined with Omega-3 in the treatment of locally advanced nasopharyngeal carcinoma.

DETAILED DESCRIPTION:
After being informed about the study and potential risks, all patients giving written informedconsent will undergo a 1-week screening period to determine eligibility for study entry. In week 0, eligible patients will be enrolled in a clinical study on the combination of Toripalimab, induction chemotherapy, sequential radiotherapy, and OMEGA-3 for the treatment of locally advanced nasopharyngeal carcinoma. Induction chemotherapy stage: Toripalimab 240mg d1, paclitaxel (albumin bound) 260mg/m2 d1, cisplatin 80mg/m2 d2 Q3W X 3 cycles. Radiotherapy stage: IMRT+Toripalimab 240mg Q3W X 3 cycles+Omega-3 (6 pills qd during radiotherapy). IMRT：GTVnx 69.96Gy，GTVnd 69.96Gy，CTV1 60Gy，CTV2 54Gy。 Maintenance treatment: Toripalimab 240mg Q3W X 6 cycles.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent can be provided, and understanding and compliance with research requirements and evaluation schedules are required.
* On the date of signing the informed consent form, the age range is between 18 and 65 years old (or the legal age specified by local laws).
* Pathological diagnosis is non keratinizing carcinoma of the nasopharynx (differentiated or undifferentiated, i.e. WHO classification II or III).
* Clinical staging is anyTN2-3M0 or T4N1M0 (AJCC8th/UICC staging).
* ECOG score is 0-1 points.
* Hemoglobin (HGB) ≥ 90g/L, white blood cell (WBC) ≥ 4.0 × 109/L, platelet (PLT) ≥ 100 × 109/L.
* Liver function: ALT and AST<2.5 times the upper limit of normal (ULN), total bilirubin<2.0 × UL, serum albumin ≥ 28g/L.
* Renal function: Serum creatinine<1.5 × ULN or creatinine clearance rate (CrCl) calculated value ≥ 60mL/min (Cockcroft Gault formula).
* Thyroid stimulating hormone (TSH) ≤ 1 × ULN (if abnormal, FT3 and FT4 levels should be examined simultaneously. If FT3 and FT4 levels are normal, they can be included in the group).
* The international normalized ratio (INR) and activated partial thromboplastin time (APTT) are ≤ 1.5 × ULN (unless the subject is receiving anticoagulant treatment and the coagulation parameters (PT/INR and APTT) are within the expected range of anticoagulant treatment at the time of screening).

Exclusion Criteria:

* Nasopharyngeal cancer patients with recurrence and distant metastasis.
* Pathology shows keratinized squamous cell carcinoma (WHO classification type I).
* Patients who have undergone radiotherapy or systemic chemotherapy before.
* Pregnant or lactating women who are in the reproductive period and have not taken effective contraceptive measures.
* HIV positive.
* Have suffered from other malignant tumors (except for cured basal cell carcinoma or cervical carcinoma in situ).
* Patients who have been treated with immune checkpoint inhibitors (CTLA-4, PD-1, PD-L1, etc.).
* Patients with immunodeficiency diseases and a history of organ transplantation.
* Patients who have been treated with high-dose corticosteroids, anti-cancer monoclonal antibodies, or other immunosuppressive agents within 4 weeks.
* Patients with significantly impaired heart, liver, lung, kidney, and bone marrow function.
* Simultaneously using other investigational drugs or in other clinical trials.
* Refusal or inability to sign the informed consent form for participation in the trial.
* Individuals with personality or mental disorders, without civil capacity or with limited civil capacity.
* hepatitis B B surface antigen (HBsAg) is positive and the peripheral blood hepatitis B virus deoxyribonucleic acid (HBV DNA) is ≥ 1000 cps/ml.
* Patients with positive HCV antibody test results are only eligible for this study if their HCV RNA polymerase chain reaction test results are negative.
* Patients who have experienced any bleeding events with a severity rating of 3 or above in CTCAE5.0 within the first 4 weeks of screening and are deemed to have a high risk of bleeding by the researchers.
* If there have been any arterial/venous thrombotic events within the 6 months prior to the start of screening, such as cerebrovascular accidents (including temporary ischemic attacks, cerebral hemorrhage, cerebral infarction), deep vein thrombosis, and pulmonary embolism.
* Patients with hypertension who cannot be reduced to the normal range through antihypertensive medication (systolic blood pressure ≥ 140mmHg or diastolic blood pressure ≥ 90mmHg); Based on the average of BP readings obtained from ≥ 2 measurements, there has been a history of hypertensive crisis or hypertensive encephalopathy.
* Past or current inflammatory bowel disease (such as Crohn's disease, ulcerative colitis, or chronic diarrhea); History of previous or existing gastrointestinal perforation and/or fistula.
* Known history of active pulmonary tuberculosis (TB). Subjects suspected of having active TB should undergo chest X-ray, sputum examination, and exclusion based on clinical symptoms and signs.
* Other serious, uncontrolled internal medical conditions and infections, or other contraindications to treatment, or any condition that researchers believe may pose a risk to receiving the study drug treatment, or interfere with the evaluation of the study drug, subject safety, or analysis of the study results.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-08-22 (Estimated); Primary Completion 2029-12-31 (Estimated); Study Completion 2029-12-31 (Estimated)

PRIMARY OUTCOMES:
2-year progression free survival period | From enrollment to the end of treatment at 2 years
  It refers to the probability of disease progression or death from any cause objectively recorded from a random date within two years, evaluated according to RECIST v1.1.

SECONDARY OUTCOMES:
objective response rate | From enrollment to the end of treatment at 2 years
  It refers to the proportion of patients who achieve complete or partial remission, evaluated by an independent review committee based on RECIST v1.1 for all randomized patients with measurable disease at baseline.
Overall survival | From enrollment to the end of treatment at 2 years
  It refers to the period from a random date to the date of death for any reason, evaluated according to RECIST v1.1.
Adverse reactions | From enrollment to the end of treatment at 2 years
  According to the National Cancer Institute's Common Terminology Criteria for Adverse Events v5.0 grading.
Quality of life score | From enrollment to the end of treatment at 2 years
  Evaluate through the European Organization for Research and Treatment of Cancer Quality of Life Questionnaire - Head and Neck Cancer-35 module and Core 30.For EORTC QLQ - H&N35:
  Title: European Organization for Research and Treatment of Cancer Quality of Life Questionnaire - Head and Neck Cancer - 35 Range: Items 1-4, subscales vary. Meaning: Higher symptom scores = worse outcome; higher functional scores (if any) = better function.
  For EORTC QLQ - C30:
  Title: European Organization for Research and Treatment of Cancer Quality of Life Questionnaire - Core 30 Range: 0-100 for scales. Meaning: Higher functional scores = better outcome; higher symptom scores = worse outcome.
  Align with standardized scoring.
Nutritional status analysis | From enrollment to the end of treatment at 2 years
  Assess nutritional status based on body mass index.Unabbreviated scale title: Body Mass Index (BMI) Minimum and maximum values: Theoretically, BMI can range from near 0 to over 100, but in practical clinical and research contexts for assessing human nutritional status, the typical relevant range is approximately 10 to 60.
  Higher scores meaning: A BMI within the normal range (18.5 - 24.9 for adults) indicates a better nutritional outcome (appropriate weight for height, supporting good health). Scores lower than 18.5 (underweight) mean a worse outcome (increased risk of nutritional deficiencies). Scores higher than 24.9 (overweight or obese, with obesity classes having higher values) also mean a worse outcome (increased risk of various health problems related to excess weight).

CONTACTS AND LOCATIONS:
Overall Officials: Haiqing Luo, doctor, Principal Investigator — Guangdong Medical University Affiliated Hospital

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data (IPD), including de - identified demographic information, clinical outcomes, and treatment details, will be shared with qualified researchers upon request. Access will be provided via a secure data repository after review and approval of a data access request form to ensure compliance with ethical and legal standards.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: IPD will become available 6 months after the primary study results are published in a peer - reviewed journal. The data will remain accessible for a period of 5 years to facilitate secondary analyses and research replication.
Access Criteria: To access IPD, researchers must: (1) Be affiliated with a recognized academic or research institution; (2) Submit a request detailing the research question, methodology, and how the data will contribute to advancing knowledge in the field; (3) Provide evidence of ethical approval from their local IRB for the proposed secondary analysis; (4) Agree to use de - identified data only and not attempt to re - identify participants. Access is granted at the discretion of the study's data governance board after a full review of the request.

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2025-06-27): https://cdn.clinicaltrials.gov/large-docs/19/NCT07136519/Prot_SAP_000.pdf
  • Informed Consent Form (2025-06-27): https://cdn.clinicaltrials.gov/large-docs/19/NCT07136519/ICF_001.pdf